CLINICAL TRIAL: NCT03801967
Title: A Phase I, Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD9977 Following Single and Multiple Ascending Dose Administration in Japanese Healthy Volunteers
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD9977 in Japanese Healthy Participants With Single and Multiple Ascending Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: D6401C00005
Record Dates: First submitted 2018-12-12; First posted 2019-01-14 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure
Keywords: Mineralocorticoid receptor; Heart failure with preserved ejection fraction; Safety; Pharmacokinetics; Single Ascending Dose; Multiple Ascending Dose
MeSH Terms: conditions — Heart Failure | interventions — AZD9977

STUDY DESIGN:
Intervention Model Description: Multiple ascending dose, placebo-controlled, single blind sequential group design
Who Masked: Participant
Masking Description: This study is single-blind (in which the study center staff have to remain blinded during the clinical conduct of a given cohort) with regard to treatment (AZD9977 or placebo) at each dose level. AZD9977 and placebo will be matched for formulation, appearance, and amount.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AZD9977 (Experimental): Each participant will receive AZD9977 at the selected dose level on Day 1 and from Day 3 to 9, with single dose on Day 1 and Day 9 and twice a day (BID) dosing on Day 3 to Day 8. No dose will be given on Day 2.
  Interventions: Drug: AZD9977
- Placebo (Placebo Comparator): Each participant will receive placebo at the selected dose level on Day 1 and from Day 3 to 9, with single dose on Day 1 and Day 9 and twice a day (BID) dosing on Day 3 to Day 8. No dose will be given on Day 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9977 — Randomized participants will receive oral dose of AZD9977.
  Arms: AZD9977
Drug: Placebo — Randomized participants will receive oral dose of matching placebo.
  Arms: Placebo

SUMMARY:
AZD9977 is an oral, selective mineralocorticoid receptor (MR) modulator. AZD9977 is a partial antagonist and partial agonist in reporter gene assays and has a different interaction pattern with the MR compared to eplerenone. This study will assess the safety, tolerability and pharmacokinetics (PK) of AZD9977, following oral administration of single and multiple ascending dose of AZD9977.

DETAILED DESCRIPTION:
This will be a Phase I, randomized, single-blind, placebo-controlled, single and multiple ascending dose sequential-group design study. The study will be conducted in healthy Japanese participants and performed at a single study center. Fourth-five healthy Japanese participants are planned to be included in the study and up to 5 additional participants may be enrolled into the study if replacement participants are needed.

Three cohorts consisting of 9 participants each will participate in the study. Depending on the findings, up to 2 additional cohorts may be added if the Safety Review Committee (SRC) considers it necessary to repeat a dose level or if additional dose steps are required.

Within each cohort, 6 participants will be randomized to receive AZD9977 and 3 participants randomized to receive placebo.

Each participant will receive AZD9977 at the selected dose level or placebo on Day 1 and from Day 3 to 9, with single dose on Day 1 and Day 9 and twice a day (BID) dosing on Day 3 to Day 8. No dose will be given on Day 2.

The study will comprise of:

* A Screening Period of maximum 28 days;
* A Treatment Period during which participants will be resident at the Clinical Unit from the day before Investigational Medicinal Product (IMP) administration (Day -1) until at least 48 hours after IMP administration; discharged on Day 11, and
* A Follow-up Visit within 5 to 7 days after the last IMP dose. Each participant will be involved in the study for approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Agree to use the methods of contraception
3. Healthy male Japanese participants aged 18 to 50 years (inclusive) with suitable veins for cannulation or repeated venipuncture. A Japanese participant is defined as having both parents and 4 grandparents who are ethnically Japanese. This includes second and third generation Japanese whose parents or grandparents are living in a country other than Japan.
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
5. Provision of signed, written and dated informed consent for optional genetic/biomarker research. If a participant decline to participate in the genetic and/or biomarker component of the study, there will be no penalty or loss of benefit to the participant. The participant will not be excluded from other aspects of the study described in this protocol.

Exclusion Criteria:

1. History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs. 3. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.

4. Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results at the Screening Visit and/or admission.

4.1. Serum potassium > 5.0 mmol/L 4.2. Hemoglobin A1c (HbA1c) > 5.7% 5. Any positive result on Screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV).

6. Abnormal vital signs, after 10 minutes supine rest at the Screening Visit and/or admission 7. Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiography (ECG) and any clinically important abnormalities in the 12 Lead ECG as judged by the Investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or LV hypertrophy at the Screening Visit and/or admission.

8. Known or suspected history of drug abuse in the last 12 months before the Screening Visit as judged by the Investigator.

9. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the previous 3 months.

10. History of alcohol abuse in the last 12 months before the Screening Visit or current excessive intake of alcohol as judged by the Investigator.

11. Positive screen for drugs of abuse, alcohol or cotinine (nicotine) at Screening or admission.

12. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD9977.

13. Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate,) as judged by the Investigator.

14. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.

15. Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, mega-dose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.

16. Plasma donation within 1 month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.

17. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit, whichever is the longest. Participants consented and screened, but not randomized in this study or a previous Phase I study, are not excluded.

18. Participants who have previously received AZD9977. 19. Involvement of any Astra Zeneca or Clinical Unit employee or their close relatives.

20. Judgment by the Investigator that the participant should not participate in the study if they have any ongoing or recent (i.e., during the Screening Period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.

21. Vulnerable participants, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

In addition, any of the following is regarded as a criterion for exclusion from the genetic research:

22. Previous bone marrow transplant. 23. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants. Serious AEs will be recorded from the time of screening.
Number of participants with abnormal blood pressure (BP) | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants. Blood pressure includes both systolic and diastolic BP.
Number of participants with abnormal supine pulse | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal findings in 12-lead safety Electrocardiogram (ECG) | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal findings in 12-lead safety Digital Electrocardiogram (dECG) | At week 5 (Visit 2)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal findings in Real-Time ECG (Cardiac Telemetry) | At week 5 (Visit 2)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal physical examination findings | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants. The complete physical examinations will include an assessment of the general appearance, skin, cardiovascular, respiratory, abdomen, head, and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Number of participants with abnormal laboratory assessments: Hematology - absolute count of Basophils, Eosinophils, Monocytes, Neutrophils, Lymphocytes and Reticulocytes; Platelets and White blood cell (WBC) count | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assesments: Hematology - Mean corpuscular volume (MCV) | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Hematology-Hematocrit (HCT) | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Hematology - Hemoglobin (Hb) | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Hematology - Red blood cell (RBC) count | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assesments: Heamtology - Mean corpuscular hemoglobin (MCH) | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assssments : Hematology - Mean corpuscular hemoglobin concentration (MCHC) | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Albumin | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Urea | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - C-reactive protein (CRP) | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Alkaline phosphatase | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Alanine aminotransferase | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Aspartate aminotransferase | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Creatinine kinase | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Creatinine | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Uric acid | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Glucose (fasting) | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Gamma glutamyl transpeptidase | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Phosphate | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Total Bilirubin and Unconjugated bilirubin | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Potassium | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Sodium | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Cholesterol | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Luteinizing hormone | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Triglycerides | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Sex hormone binding globulin | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Follicle-stimulating hormone | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Testosterone | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Aldosterone | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Hemoglobin A1c | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Clinical Chemistry - Electrolytes | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants. Electrolyte Measurements includes Bicarbonate, Calcium, Chloride, Potassium, Sodium
Number of participants with abnormal laboratory assessments: Clinical Chemistry - High-sensitive-CRP | At Visit 2 (Week 5)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: High-sensitivity Troponin T | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: N-terminal pro-brain Natriuretic Peptide | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal urine volume | At Visit 2 (Week 5)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Urinalysis - Glucose | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Urinalysis - Protein | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants.
Number of participants with abnormal laboratory assessments: Urinalysis - Blood | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants. Microscopy should be done (if positive for protein or blood): red blood cells (RBC), white blood cells (WBC), Casts (Cellular, Granular, Hyaline)
Number of participants with abnorml laboratory assessments: Urinalysis - Urinary Electrolytes | From screening (Day -28) till follow-up visit (Up to 6 weeks)
  To investigate the safety and tolerability of AZD9977 following oral administration of single and multiple ascending doses at steady state in healthy Japanese participants. Urinary Electrolytes: Calcium, Potassium, Chloride, Sodium, Creatinine and Uric acid.

SECONDARY OUTCOMES:
Plasma PK analysis: Area under curve (AUC) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Maximum observed plasma concentration (Cmax) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Time to reach peak or maximum observed concentration following drug administration (tmax) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Observed concentration at the end of the dosing interval following drug administration (Cmin) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Terminal elimination rate constant, estimated by log-linear least squares regression of the terminal part of the concentration-time curve following drug administration (λz) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Terminal half-life, estimated as (ln2)/λz (t½λz) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Area under the plasma concentration-time curve from time zero to the time of the last measurable concentration (AUClast) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Area under the plasma concentration-time curve in the dosing interval (AUCτ) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Renal clearance, estimated by dividing Amount of analyte excreted into the urine(0-t) [Ae(0-t)] by AUC(0-t) where the time interval for both parameters are the same (CLr) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Mean Residence Time (MRT) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Apparent volume of distribution for parent drug at terminal phase, estimated by dividing the apparent clearance (CL) by λz (Vz/F) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Area under the plasma concentration-time curve from time zero extrapolated to infinity divided by the dose administered (AUC/D) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Area under the plasma concentration-time curve from time zero to the time of the last measurable concentration divided by the dose administered (AUClast/D) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Area under the plasma concentration-time curve in the dosing interval divided by the dose administered (AUCτ/D) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Observed maximum plasma concentration divided by the dose administered (Cmax/D) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Accumulation ratio for AUCτ, estimated by dividing AUCτ from the last dosing day by AUCτ on Day 1 (Rac AUCτ) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Accumulation ratio for Cmax (Rac Cmax) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Plasma PK analysis: Temporal change, estimated by dividing AUCτ from the last dosing day by AUC on Day 1 (TCP) | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Urine PK analysis: Amount of analyte excreted into the urine from time t1 to t2 [Ae(t1-t2)] | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.
Urine PK analysis: Percentage Fraction of dose excreted in urine from time t1 to t2, estimated by dividing Ae(t1-t2) by dose * 100 [fe(t1-t2)%] | Day 1-2: Pre-dose and 0-4, 4-8, 8-12 and 12-24 hours post-dose and Day 9: Pre-dose and 0-4, 4-8 and 8-12 hours post-dose
  To characterize the single and multiple dose PK of AZD9977 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK in healthy Japanese participants.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Forte Soto, MD, MSc, PhD, Principal Investigator — Dr
Locations (1):
- Research Site, Harrow, United Kingdom